CLINICAL TRIAL: NCT05264623
Title: A Study to Investigate the Safety and Effectiveness of the TENEO 317 Model 2 (1.28 US) Excimer Laser for Laser In Situ Keratomileusis (LASIK) Surgery to Treat Hyperopia With or Without Astigmatism
Brief Title: Safety and Effectiveness of the TENEO 317 Model 2 (1.28 US) Excimer Laser for Laser In Situ Keratomileusis (LASIK) Surgery to Treat Hyperopia With or Without Astigmatism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 906
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hyperopia
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- TENEO 317 Model 2 excimer laser (Experimental)
  Interventions: Device: TENEO 317 Model 2 excimer laser

INTERVENTIONS:
Device: TENEO 317 Model 2 excimer laser — TENEO 317 Model 2 excimer laser use for refractive surgery

SUMMARY:
This will be a multicenter, prospective, open label, non-randomized, single arm 12 month study, evaluating the safety and effectiveness of the TECHNOLAS TENEO 317 Model 2 (Software version "1.28 US") excimer laser when used in LASIK surgery to treat hyperopia with or without hyperopic astigmatism. Both eyes of a subject may be enrolled so long as both eyes meet all inclusion/exclusion requirements. Analysis of the primary effectiveness endpoint will be completed at refractive stability.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 22 years of age or older at the time of the pre-operative examination.
2. Manifest, distance corrected visual acuity (CDVA) 20/25 (logMAR 0.10) or better in an operative eye
3. Pre-operative refractive error of hyperopia with spherical component of 0.00 D to +4.00 D with or without cylinder up to +2.00 D, with MRSE of ≥ 0.375 D and ≤ +5.00 D based on the manifest refraction in thestudy eye(s). This would exclude eyes with cylinder-only corrections < +0.75D and sphere-only corrections < +0.375D)
4. Difficulty maintaining uncorrected distance visual acuity (UDVA) of 20/40 or better, as evidenced by need for constant contact lens or spectacle wear.
5. Difference between manifest refractive and cycloplegic spherical equivalent ≤ 0.75 D, difference between manifest and cycloplegic cylinder ≤ ± 0.50 D and difference between manifest and cycloplegic cylinder axis ≤ ± 15 degrees.
6. Stable refraction (i.e., a change of ≤ ± 0.50 D in MRSE) for a minimum of 12 months prior to surgery, as verified by consecutive refractions, medical records, or prescription history.
7. Agree to discontinue use of contact lenses for at least 2 weeks (for rigid or toric lenses) or 3 days (for soft contact lenses) prior to the first refraction used to establish stability and through the day of surgery.
8. All contact lens wearers must demonstrate a stable refraction in an eye to be treated, as follows: two consecutive examinations at least 1 week apart within ± 0.50 D manifest refractive spherical equivalent and within ± 15 degrees cylinder axis.
9. Agree to emmetropia correction for each treated eye.
10. Anticipated postoperative stromal bed thickness of at least 250 microns.
11. Can lie flat without difficulty.
12. Willing and able to read, understand, and sign a written informed consent form (ICF).
13. Willing and able to comply with the schedule for all post-surgery follow-up visits.

Exclusion Criteria:

1. Acute or chronic disease or illness that would increase operative risk or confound the results of the study (e.g., dry eye disease, cataract, glaucoma, immuno-compromised, rheumatoid arthritis, clinically significant atopic disease, acne rosacea, autoimmune disease, endocrine disorders, lupus, systemic connective tissue disease, diabetes, or severe atopic disease).
2. Use of medications by any administration route that may increase risk to the subject or may confound the outcome of the study, including those known to affect wound healing (e.g., systemic corticosteroids, antimetabolites).
3. Ocular conditions, other than hyperopia with or without astigmatism that may predispose the subject to future complications including but not limited to:

   1. Evidence or history of retinal vascular disease
   2. Evidence or history of active or inactive corneal disease or infection (e.g., recurrent corneal erosion syndrome, herpes simplex or herpes zoster keratitis) in either eye.
   3. Evidence or history of glaucoma or glaucoma suspect (IOP > 24mmHg) by exam findings and/or family history
4. Previous intraocular or corneal surgery in an eye considered for eligibility that might confound the outcome of the study or increase the risk to the subject.
5. An increased risk for developing strabismus post-treatment or an ocular muscle disorder (e.g., strabismus or nystagmus) affecting fixation.
6. Known sensitivity to any study medications (e.g., used during LASIK procedure and postoperative care).
7. Have central corneal scars affecting visual acuity.
8. Have mixed astigmatism.
9. Presence of keratoconus, keratoconus suspect, subclinical or forme fruste keratoconus, corneal dystrophy, or other corneal irregularity (e.g., irregular astigmatism) or abnormal corneal topography
10. Presence of visually significant or progressive cataract in an eye considered for eligibility.
11. Actively taking medications contraindicated with LASIK such as isotretinoin (Accutane) or amiodarone hydrochloride (Cordarone).
12. Have a cardiac pacemaker, implanted defibrillator, or other implanted electronic device.
13. Pregnant, lactating, or subjects who plan to become pregnant during the course of the study.
14. Are participating in any other trial within 30 days of screening or during this clinical trial.
15. Eyes with mesopic pupil size > 7.0 mm.
16. Have a Schirmer's pre-operative test without anesthesia < 4 mm after 5 minutes

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
The percentage of eyes with Uncorrected Distance Visual Acuity (UDVA) of 20/40 or better at the time of refractive stability | Up to 12 months
The percentage of eyes with Manifest Refractive Spherical Equivalent (MRSE) within 0.50 Diopter of intended correction at the time of refractive stability | Up to 12 months
The percentage of eyes with Manifest Refractive Spherical Equivalent (MRSE) within 1.00 Diopter of intended correction at the time of refractive stability | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosangela Nolasco, Study Director — Bausch & Lomb Incorporated
Locations (9):
- United States (9):
  - Site 113, Newport Beach, California
  - Site 111, Fort Myers, Florida
  - Site 101, Bloomington, Minnesota
  - Site 104, Saint Louis Park, Minnesota
  - Site 103, Omaha, Nebraska
  - Site 102, Amherst, New York
  - Site 112, Pittsburgh, Pennsylvania
  - Site 108, Sioux Falls, South Dakota
  - Site 106, Cedar Park, Texas

IPD SHARING:
Plan to Share IPD: Undecided